CLINICAL TRIAL: NCT05855824
Title: Controlled Trial to Validate Skin Carotenoid Dietary Biomarker in Toddlers
Brief Title: Toddler Biomarker of Nutrition Study
Acronym: TBONS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: University of Houston (Other); East Carolina University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Nancy Engelmann Moran, Assistant Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: H-53006; 1R01HD111555 (NIH)
Record Dates: First submitted 2023-04-25; First posted 2023-05-12 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Pediatric Nutrition; Nutrition, Healthy
Keywords: carotenoids; nutritional biomarkers; nutrition assessment; pediatric nutrition; skin carotenoids; fruits and vegetables
MeSH Terms: interventions — Mangifera indica extract

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to a low, medium, or high carotenoid food intervention.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator and statisticians on the team will be blinded. A staff member outside of the team will be responsible for randomly assigning and dispensing the study foods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo - 0 mg carotenoids / d (Placebo Comparator): The placebo "0 mg/d" group consumes 1-90 g pouch of applesauce providing 0 mg carotenoids/d (Unsweetened Applesauce Pouches) daily for 4 weeks.
  Interventions: Other: Applesauce Pouch
- Low - 2.5 mg carotenoids / d (Experimental): The low "2.5 mg/d" group will consume alternating pouches of the applesauce (0 mg carotenoids/90 g pouch) and a 120 g pouch of fruit-vegetable puree blend providing 5 mg mixed carotenoids (Carrot, Banana, Mango, & Sweet Potato pouch) daily for 4 weeks.
  Interventions: Other: Applesauce Pouch; Other: Fruit-vegetable puree blend
- High - 5 mg carotenoids / d (Experimental): The high dose "5 mg/d" group will be provided one 120 g pouch/day of the fruit-vegetable puree blend (Carrot, Banana, Mango, & Sweet Potato pouch) daily for 4 weeks.
  Interventions: Other: Fruit-vegetable puree blend

INTERVENTIONS:
Other: Applesauce Pouch — One 90 g pouch of applesauce provides 0 mg carotenoids/d and 40 kcal, 10 mg vitamin C, and 1 g dietary fiber.
  Other Names: Unsweetened Applesauce Pouches, Mott's Inc.
  Arms: Low - 2.5 mg carotenoids / d; Placebo - 0 mg carotenoids / d
Other: Fruit-vegetable puree blend — One 120 g pouch of fruit-vegetable puree blend provides 5 mg mixed carotenoids, 70 kcal, 4 mg vitamin C, and 2 g dietary fiber.
  Other Names: Carrot, Banana, Mango, & Sweet Potato pouch, Happy Tot, Happy Family Brands
  Arms: High - 5 mg carotenoids / d; Low - 2.5 mg carotenoids / d

SUMMARY:
This is a study of how accurate different methods to assess young children's dietary intake are, so that researchers and health professionals can better understand how children's nutrition relates to their health. The study will compare food surveys, measurements of nutrients in the blood, and optical measurements of nutrients in the skin.

DETAILED DESCRIPTION:
Young children rely on their foods and drinks for the nutrients they need to grow, like energy, protein, vitamins, and minerals. However, it is challenging for researchers to study children's nutrition, because it is difficult to rapidly and accurately assess what exactly children eat. This is a study of different methods to assess young children's dietary intake so that researchers can better understand how children's nutrition relates to their health. The study will compare food surveys, measurements of nutrients in the blood, and optical measurements of nutrients in the skin to see how well these different measures agree with one another.

Carotenoids are a group of natural red, orange, and yellow substances found in fruits and vegetables. Children and adults absorb carotenoids from their foods. Measurements of the amounts of carotenoids in blood or optically in the skin can serve as to indirectly measure what a person eats. Optical skin carotenoid measurements could be a simple alternative to blood sampling or dietary surveys for researchers and practitioners in medicine and public health to quickly assess children's diets. What is unknown is how long it takes for blood or skin carotenoid measurements in young children to change in response to a change in their diet. Also, how accurately the blood and skin carotenoid measurements reflect the changes in a child's diet is unknown.

For this research study, volunteers to report on what their child eats over the course of 4 weeks. Participants will also incorporate specific fruit and/or fruit and vegetable blended puree pouches into their toddler's daily eating pattern. The study will follow how quickly the skin and blood measurements change in response to specific changes to the child participant's eating patterns. The study involves 3 visits and consuming a study-provided food every day for 4 weeks. At each visit, parents will report on the participating child's recent eating pattern, the study team will measure the child participant's body size and skin fold thicknesses as a measure of body composition, collect a blood sample (1 teaspoon), and do optical measurements of their skin. At visit 1, child participants will be randomly assigned to consume a daily applesauce pouch, or a carrot-mango-banana-sweet potato pouch, or alternate between the two pouches, for the next 4 weeks. The adult guardian and the child participants then return at 14 and 28 days. Before the last two visits, the adult participant will complete online surveys about what their child has been eating.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* 24 months of age
* categorized by their guardian caregiver as either non-Hispanic white, Asian, Hispanic white, or non-Hispanic Black
* participating guardian speaks, reads, and understands English.

Exclusion Criteria:

* metabolic, endocrine, or digestive condition, food intolerance, or food allergy
* bleeding or clotting disorder
* taking a medication or complementary alternative medicine that would interfere with fat absorption
* taking a dietary supplement that provided more than 1 mg carotenoids per day
* has a sibling that is participating or participated in the study.

Ages: 24 Months to 26 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline skin carotenoid concentration at 4 weeks | Four weeks
  Change in pressure mediated reflection spectroscopy measurement of total carotenoids at the finger over 4 weeks.

SECONDARY OUTCOMES:
Change from baseline serum carotenoid concentration at 4 weeks | Four weeks
  Total plasma carotenoids (sum of beta-carotene, alpha-carotene, lutein, zeaxanthin, lycopene, and beta-cryptoxanthin) in participant plasma.

OTHER OUTCOMES:
Change from baseline dietary carotenoid intake at 4 weeks | Four weeks
  Dietary carotenoid intake assessed by 3-day food diary
Intervention adherence | Daily from baseline to end of study (4 weeks)
  Amount of the intervention foods consumed daily, recorded by adult guardians.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy E. Moran, PhD, Principal Investigator — Baylor College of Medicine

IPD SHARING:
Plan to Share IPD: No